CLINICAL TRIAL: NCT03830762
Title: XanaHES: A Phase I, Single Blinded, Central Reader Blinded, Placebo-Controlled, Dose Escalation Study of Xanamem™ to Assess Safety and Tolerability in Healthy Elderly Subjects
Brief Title: Xanamem™ in Healthy Elderly Subjects
Acronym: XanaHES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actinogen Medical (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ACW0003
Record Dates: First submitted 2019-01-23; First posted 2019-02-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2020-08

CONDITIONS: Safety; Peripheral Neuropathy; Cortisol; Central Nervous System; Cognitive Function; Healthy Ageing; Small Fibre Neuropathy; Cerebrospinal Fluid; Electrocardiography
Keywords: Actinogen; Xanamem; UE2343; Cortisol; 11β-HSD1; 11-beta-Hydroxysteroid Dehydrogenase Type 1; Healthy Ageing; Peripheral Neuropathy; Safety; Dose Escalation; Elderly; XanaHES; emestedastat
MeSH Terms: conditions — Peripheral Nervous System Diseases; Small Fiber Neuropathy | interventions — UE2343

STUDY DESIGN:
Intervention Model Description: A Dose Escalation Committee will review the results from Cohort 1 (20 mg active vs. placebo arms) and provide a recommendation to proceed with Cohort 2 (30 mg active vs. placebo arms) randomisation which involves a dose escalation.
Who Masked: Participant
Masking Description: Study treatment is only blinded for the trial subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 / Cohort 2 (Active) (Experimental): 20mg or 30mg capsules of Xanamem respectively, to be administered PO once daily.
  Interventions: Drug: Xanamem
- Cohort 1 / Cohort 2 (Placebo) (Placebo Comparator): Matching placebo which is identical in appearance to the test product except that it contains no active ingredient, to be administered once daily.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Xanamem — Oral Xanamem capsules 20mg or 30mg, administered PO once daily. Xanamem is formulated in green and cream coloured size 3, Coni-Snap shaped gelatin capsules as an excipient blend at a dose of 10mg. It contains active pharmaceutical ingredient of UE2343.
  Other Names: UE2343
  Arms: Cohort 1 / Cohort 2 (Active)
Drug: Matching Placebo — Matching placebo which is identical in appearance to the test product (20mg, 30mg Xanamem™ QD) except that it contains no active ingredient.
  Other Names: Placebo
  Arms: Cohort 1 / Cohort 2 (Placebo)

SUMMARY:
Xanamem™ is being developed as a potential drug for Alzheimer's disease. This study drug has been designed to change the cortisol levels in the brain. Cortisol is a naturally occurring hormone in the body. It is believed that reducing the level of cortisol will be a benefit in the treatment of Alzheimer's disease.

The XanaHES study is testing the safety and tolerability of Xanamem. It is planned to enrol approximately 84 participants, male and female aged from 50 to 75 who are in good health, in the study at 1 centre in Australia.

The XanaHES Phase I study is a single-blind study. Subjects will be randomised to receive either 20mg once daily Xanamem or Placebo in cohort 1. Once all subjects have completed the study treatment of 12 weeks, a dose escalation committee will decide if a new cohort, cohort 2, with 30mg once daily vs placebo is started.

DETAILED DESCRIPTION:
This is a Phase I, randomised, single-centre, single-blind, placebo-controlled study to assess the safety, tolerability of oral Xanamem once daily in healthy elderly subjects.

It is planned to randomise approximately 84 subjects, 42 in each cohort, at a single site in Australia.

Cohort 1 starts with a 20mg QD dose vs matching placebo. A Dose Escalation Committee will review the results from cohort 1 and provide a recommendation to proceed with Cohort 2 randomisation which involves a dose escalation to 30mg.

At the Baseline visit (Week 0), eligible subjects will be randomised on a 30:12 ratio to receive either Xanamem administered orally QD (treatment group) or matching placebo (placebo group). Subjects will return to the study site for visits at Week 2, Week 4, Week 6, Week 8, Week 10, End of Treatment (Week 12) and Follow-up (4 weeks post last dose of study drug) visits, at which study assessments will be performed.

Ad hoc telephone contact may also occur at any other time-point throughout the study, if deemed necessary by the investigator/study nurse, or if the subject wishes to report an adverse event (AE).

Subjects will be interviewed and examined at the study site at each visit and will complete a variety of questionnaires, routine safety evaluations and nerve function tests.

A central reader will review every Nerve Function Monitoring (NFM) assessment performed for each subject for Potential Nerve Safety Signals (PNSS).

Optional cerebrospinal fluid (CSF) sampling will be performed at baseline and end of treatment visits for a small subgroup of subjects, who provide additional consent. Subjects who do not provide consent for this optional sub-study will still be eligible for the main study.

The overall study duration for an individual subject will be 17 to 20 weeks, including a screening period of up to 4 weeks, a single-blind treatment period of 12 weeks, and a follow-up period of 4 weeks. The total duration of the study is expected to be 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 50 to 75 years.
2. Female subjects:

   1. Post-menopausal women, defined as no menses for 12 months without an alternative medical cause. If there is any concern about the menopausal status of a prospective female subject, a follicle stimulating hormone test (FSH) should be requested to confirm post-menopausal status. Post-menopausal women confirmed by FSH level > 40 mIU/mL, will be confirmed by the local laboratory.
   2. Women of childbearing potential (WOCBP) must have a negative pregnancy test.
3. Male Subjects:

   1. Who are sexually active, fertile men must use highly effective methods of contraception from Day 1 until 3 months after last dose of study drug if their partners are WOCBP
   2. Who are permanently sterile or have had bilateral orchiectomy or bilateral vasectomy.
4. No disease which may cause a peripheral neuropathy.
5. No evidence of alcohol abuse (defined as greater than 21 standard units per week for males and greater than 14 standard units per week for females).
6. Must provide written informed consent to participate in the study and be willing and able to participate for the maximum of 12 weeks of treatment and 16 weeks of site visits.

Exclusion Criteria:

1. Clinically significant abnormalities in vital signs (blood pressure, heart rate, respiration rate and oral temperature), as determined by the investigator.
2. Body Mass Index (BMI) > 38 kg/m2
3. Clinically significant abnormal haematology, biochemistry and urine examination values, as determined by the investigator.
4. Participants who have a history of liver disease, including fatty liver, or LFT elevations requiring investigation will not be eligible.
5. Has had a significant systemic illness or infection within the past 4 weeks prior to randomisation, as determined by the investigator.
6. Documented diagnosis of Type I or Type II diabetes.
7. Has a history of disease directly related to the hypothalamus, the pituitary and/or the adrenal glands which affects the hypothalamic-pituitary-adrenal axis function.
8. Has any uncontrolled clinical condition relating to glucose or lipid metabolism.
9. Subjects with clinical evidence of peripheral neuropathy or historical evidence of clinically significant nerve conduction abnormalities. Clinical evidence of neuropathy.
10. Clinically significant electrocardiogram (ECG) abnormalities, including QTc interval > 450 msec (male) and > 470 msec (female), following ECG tracings at Screening.
11. Use of any prohibited medication.
12. Participation in another clinical study of a drug or device whereby the last investigational drug/device administration is within 60 days of Screening.
13. Inability to communicate well with the investigator (i.e. language problem, non-fluent English [as questionnaires and study drug label will be provided in English only], poor mental development or impaired cerebral function).
14. Subject will undergo the Columbia Suicide Severity Rating Scale (CSSRS), Toronto Clinical Neuropathy Score (TCNS), EuroQoL Health Related Quality of Life - 5 Dimensions - 5 Levels (EQ-5D-5L), and Cogstate Test Battery at the indicated time-points to avoid uncontrolled learning effects. Subjects who need to perform these tests externally to and in parallel with this study will be excluded.
15. For subjects that consent, and are subsequently accepted for enrolled into, the CSF optional sub-study, subjects must have no contraindications to the lumbar puncture procedure as assessed by the Principal Investigator. Such contraindications may include uncontrolled bleeding abnormalities or skin or spine abnormalities.
16. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV). Subjects returning a positive result will be managed by the site in line with standard care.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) | 20 Weeks (Screening up to Week 16 Follow-Up [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  The number, type, and severity of treatment-emergent adverse events (AEs) that are reported from Screening Visit to Follow-up Visit will be collected and evaluated.
Incidence of Clinically Significant Changes in Serum Biomarker Levels in a Standard Serum Chemistry Panel | Screening up to Week 16 (Follow-Up [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Collection of blood samples for clinical laboratory testing to assess any clinically significant changes in standard serum chemistry measures.
Incidence of Clinically Significant Laboratory Haematological Biomarker Levels in a Standard Haematology Panel. | Screening up to Week 16 (Follow-Up [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Collection of blood samples for clinical laboratory testing to assess any clinically significant changes in standard haematology measures.
Incidence of Clinically Significant Changes or Abnormalities Following Physical Examination | Screening up to Week 16 (Follow-Up) and Unscheduled Safety Visit throughout duration of study up to Week 16 (Follow-Up Visit [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Evaluation of any clinically significant changes or abnormalities reported following a standard Physical Examination.
Nerve Conduction Assessments | Screening up to Week 16 (Follow-Up Visit [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Nerve Conduction assessments will be used to detect presence and severity of nerve damage.
Neuropathy Total Symptom Score-6 (NTSS-6) | Screening, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up) and Telephone Contact (Ad Hoc)
  Changes in the Neuropathy Total Symptom Score (NTSS-6) administered by a physician to assess a subjects' medical history. Each item will also be graded for its frequency and intensity, adding up to a total score from "0" to "21.96" points. A total score of > 6 would exclude the subject from the study.
Toronto Clinical Neuropathy Score (TCNS) | Screening, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up) and Telephone Contact (Ad Hoc)
  Changes in Toronto Clinical Neuropathy Score (TCNS) to detect for neuropathy out of a total score of 19; scales are defined as follows: 0-5 = no neuropathy; 6-8 = mild neuropathy; 9-11 = moderate neuropathy; ≥ 12 = severe neuropathy.
Skin Biopsy | At Baseline and Week 12 (End of Treatment)
  A 3mm skin sample will be taken via skin punch biopsy to detect intra-epidermal nerve fiber density; this allows for the objectification and quantification of a small-fiber neuropathy.
Quantitative Sensory Testing (QST) | Screening up to Week 16 (Follow-Up Visit [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Thermal sensory testing using Quantitative Sensory Testing (QST) for cold, warm and heat pain to detect peripheral nerve disorders.
Columbia Suicide Severity Rating Scale (CSSRS) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Any change in Columbia Suicide Severity Rating Scale (CSSRS) will assess suicidal ideation and behaviour.
  * Suicidal ideation score: Any score greater than 0 is important and may indicate the need for mental health intervention.
  * Suicidal ideation intensity rating: The five intensity item scores create a total score (range 0 to 25) to represent the intensity rating, if the patient did not endorse any suicidal ideation the intensity rating is 0.
Electrocardiogram (ECG) | Screening up to Week 16 (Follow-Up Visit [4 Weeks Post Last Dose of Study Drug ± 4 Days])
  Any clinically significant electrocardiogram (ECG) abnormalities will be recorded, including corrected QT interval (QTc) of > 500 msec.

OTHER OUTCOMES:
Detection Test (Cogstate Test Battery) | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Changes in Cogstate Detection test is a measure of simple reaction time and has been shown to provide a valid assessment of psychomotor function. For this test, the subject must press a "YES" response key as soon as they detect an event (i.e. a card turning face up presented in the centre of the computer screen). The software measures the response time to detect each event.
Identification Test (Cogstate Test Battery) | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Changes in the Cogstate Identification test is a measure of choice reaction time and has been shown to provide a valid assessment of visual attention. In this test an event (a card turning face up) occurs in the centre of the computer screen and the subject must decide "YES" or "NO" as to whether this event meets a predefined and unchanging criterion (is the colour of the card red?). The software measures the speed and accuracy of each response.
One Back Working Memory Test (Cogstate Test Battery) | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Changes in Cogstate the Cogstate One Back memory test is a valid measure of working memory. On this test the subject is shown a single stimulus in the centre of the computer screen (a card turns face up). They must decide "YES" or "NO" as to whether the current card matches the card that had been seen on the immediately previous trial. The software measures the speed and accuracy of each response.
One Card Learning Test (Cogstate Test Battery) | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Changes in Cogstate the One Card Learning test is a continuous visual recognition learning test that assesses visual learning within a pattern separation model. The One Card Learning test has been shown to be a valid test of learning and memory. In this test the participant must attend to the card in the centre of the screen and respond to the question "have you seen this card before in this test?" If the answer was yes, participants are instructed to press the "YES" button, and the "NO" button if the answer is no. Normal playing cards are displayed (without joker cards). In this test, six cards are drawn at random from the deck and are repeated throughout the test. These four cards are interspersed with distractors (non-repeating cards). The test ends after 50 trials, without rescheduling for post-anticipatory correct trials. The primary performance measure for this test is the proportion of correct answers (accuracy), which is normalized using an arcsine square root transformation.
Continuous Paired Associate Learning Test ([CPAL; Paired Associate Learning] Cogstate Test Battery) | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up)
  Changes in Cogstate the Continuous Paired Associate Learning test is a measure of visual associate memory and uses a well-validated paired associate learning paradigm in which the subject must learn the locations of a number of amoeba-like shapes on the computer screen. Finding the correct location for all patterns in the set is defined as a learning trial. There are six learning trials. A single trial delayed recall condition is available for this test after a 10-30-minute delay. The software records each move as an error or as a correct move.
Pharmacokinetics Blood Sample Assessment | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment), Week 16 (Follow-Up) and Unscheduled Safety Visit throughout duration of study up to Follow-Up Visit (4 Weeks Post Last Dose of Study Drug ± 4 Days)]
  Changes in area under the plasma concentration versus time curve (AUC). Peripheral pharmacokinetic (PK) blood samples will be taken from all enrolled subjects.
Cortisol Concentration | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment) and Week 16 (Follow-Up)
  Changes in peripheral cortisol concentration levels with analysis of Pharmacokinetics (PK) blood samples.
Optional Cerebrospinal Fluid Assessment | Week 12 (End of Treatment)
  An optional CSF assessment will be offered to willing participants to detect changes in CSF levels from a minimum of 8 enrolled subjects, 4 subjects from each cohort, randomised to active treatment, for those who consent to take part in the CSF sub-study. Two CSF samples will be taken End of Treatment (EOT) at Week 12 visit, one for primary analysis and one sample to be retained for back-up purposes.
Health Related Quality of Life: EQ-5D-5L | Baseline, Week 2, Week 4, Week 8, Week 12 (End of Treatment) and Week 16 (Follow-Up)
  Overall Health Related Quality of Life (HRQoL) will be assessed by EuroQoL Health Related Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L). The EQ-5D-5L is a standardized, participant-rated questionnaire for use as a measure of health outcomes.
  The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the visual analogue scale (VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
  For each dimension, the participant is instructed to choose one of 5 levels that best describes their health on that day: "no problem" (1), "slight" (2), "moderate" (3), "severe" (4), or "unable/extreme" (5). The VAS is the participant's rating of their health on a scale of 0 "worst health you can imagine" to 100 "best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Bill Ketelbey, MD, Study Chair — Actinogen Medical
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webster SP, McBride A, Binnie M, Sooy K, Seckl JR, Andrew R, Pallin TD, Hunt HJ, Perrior TR, Ruffles VS, Ketelbey JW, Boyd A, Walker BR. Selection and early clinical evaluation of the brain-penetrant 11beta-hydroxysteroid dehydrogenase type 1 (11beta-HSD1) inhibitor UE2343 (Xanamem). Br J Pharmacol. 2017 Mar;174(5):396-408. doi: 10.1111/bph.13699. Epub 2017 Jan 25. PMID 28012176